CLINICAL TRIAL: NCT00447512
Title: Effects of Ghrelin on the Sleep-EEG and Nocturnal Secretion of Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: L2/2003
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Healthy; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ghrelin — acylated ghrelin

SUMMARY:
Ghrelin, an acylated peptide consisting of 28 amino acids, is the endogenous ligand of the growth hormone secretagogue receptor (GHS-R). It is synthesized predominantly in the stomach but has been also identified in a variety of other organs. Alike, a wide range of central and peripheral endocrine and non-endocrine actions has been described, e. g. being a releasing factor of growth hormone, prolactin and ACTH, a modulator of cell proliferation and apoptosis, a regulator of sleep-wake regulation, and a orexigenic hormone. Aims of this study are:

A) To determine the effect of exogenous ghrelin on sleep-EEG variables and hormones of the hypothalamic-pituitary-adrenocortical (HPA) axis, the gonadotropic axis and the hypothalamic-pituitary-gonadal axis in healthy subjects of both genders (age groups: 20-30, 35-45, 60-70 years).

B) To determine the effect of exogenous ghrelin on sleep-EEG variables and hormones of the HPA axis, the gonadotropic axis and the hypothalamic-pituitary-gonadal axis in patients with major depression (age range: 20-65 years).

ELIGIBILITY:
Inclusion Criteria:

* Healthy females and males
* Male and female patients with major depression

Exclusion Criteria:

* Life time or family history of psychiatric or neurological disorders
* Sleep disturbances
* Shift work
* Any current disease
* Any medication
* Long distance flight within 3 months prior to study entry
* Smoking
* Any medication during the week prior to study entry
* Any current disease other than major depression

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
sleep, conventionally and quantitatively analyzed | study duration

SECONDARY OUTCOMES:
hormones of the hypothalamic-pituitary-adrenocortical (HPA) axis, the gonadotropic axis and the hypothalamic-pituitary-gonadal axis | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Professor Axel Steiger, MD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Germany

REFERENCES:
- [Derived] Kluge M, Schussler P, Schmidt D, Uhr M, Steiger A. Ghrelin suppresses secretion of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) in women. J Clin Endocrinol Metab. 2012 Mar;97(3):E448-51. doi: 10.1210/jc.2011-2607. Epub 2012 Jan 18. PMID 22259063